CLINICAL TRIAL: NCT03941522
Title: Loop Ileostomy Closure as a 23-hour Stay Procedure, a Multi-center Randomized Controlled Trial
Acronym: ILEO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CHU de Quebec-Universite Laval (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019-4382
Record Dates: First submitted 2019-05-06; First posted 2019-05-08 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Ileostomy - Stoma
Keywords: loop ileostomy; diversion ileostomy; ileostomy closure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (23-hour stay) (Experimental): Patients randomized to the group 23-hour stay will be discharged on the day after their surgery if they meet the discharge criteria.
  Interventions: Other: Early discharge from hospital
- Control group (conventional hospitalization) (No Intervention): Patients randomized to the group conventional hospitalization will be hospitalized as per the current conventional care after ileostomy closure.

INTERVENTIONS:
Other: Early discharge from hospital — Patients randomized to the group 23-hour stay will be discharged on the day after their surgery if they meet the discharge criteria.
  Arms: Intervention group (23-hour stay)

SUMMARY:
The purpose of this study is to assess the safety and feasibility of ileostomy closure performed in a 23 hours hospitalization setting, using a multi-center, open-label, randomized controlled trial comparing patients being hospitalized overnight (discharged on the day after surgery) to patients being hospitalized as per the current conventional care after ileostomy closure with both groups following a standardized enhanced recovery after surgery (ERAS) pathway specific to ileostomy closure. Primary outcome will be total length of hospital stay in days and secondary outcomes, measured at 30 days, will include readmission rate, postoperative complication rate minor and severe, postoperative ileus rate, postoperative surgical site infection rate and mortality rate.

DETAILED DESCRIPTION:
Rationale :

Loop ileostomy is defined by bringing a loop of small bowel out onto the surface of the skin to allow diversion of the fecal stream. It is a common procedure that is conjointly done with colorectal surgeries with the objective to protect intestinal anastomosis at high risk of leaking. Loop ileostomy closure is then performed in the months following the initial surgery when the anastomosis has healed. Often thought of as a simple procedure, it is still associated with a significant postoperative morbidity rate consisting mostly of postoperative ileus. In the CHU de Québec-Université Laval, patients are hospitalized for a median of five days until their bowels open up while no active care is given. This represents 645 days of hospitalization each year for Hôpital Saint-François d'Assise (HSFA), Hôtel-Dieu de Québec (HDQ) and Centre Hospitalier de l'Université Laval (CHUL). Hence, there is a clear need to determine if the investigator can improve the outcomes following ileostomy closure by applying a standardized enhanced recovery pathway specific to ileostomy closure to the point where the surgery can be performed in a twenty-three hours hospitalization setting.

Objective :

The purpose of this study is to assess the safety and feasibility of ileostomy closure performed in a 23 hours hospitalization setting, using a multi-center, open-label, randomized controlled trial comparing patients being hospitalized overnight (discharged on the day after surgery) to patients being hospitalized as per the current conventional care after ileostomy closure with both groups following a standardized enhanced recovery after surgery (ERAS) pathway specific to ileostomy closure. Primary outcome will be total length of hospital stay in days and secondary outcomes, measured at 30 days, will include readmission rate, postoperative complication rate minor and severe, postoperative ileus rate, postoperative surgical site infection rate and mortality rate.

Hypothesis :

The investigator believes patients randomized to the group 23-hour stay will have reduced total length of hospital stay compared to patients randomized to the group conventional hospitalization after ileostomy closure.

Methods :

Healthy adults (ASA I and II) undergoing elective ileostomy closure who consented to take part in the study will be enrolled in a standardized enhanced recovery pathway specific to ileostomy closure. Once surgery is completed, they will be randomized to either 23-hour stay or conventional hospitalization. Data on postoperative outcomes will be gathered prospectively until 30 days after surgery and will include total length of hospital stay in days, readmissions, postoperative complications, more precisely postoperative ileus and surgical site infections, as well as mortality.

Clinical significance :

If safety and feasibility of a fast discharge of patients is demonstrated by this study, it would then mean that patients could be discharged from hospital less than 24 hours after a loop ileostomy closure. It could potentially lower the consequences of a long hospital stay for patients, such as risks of nosocomial infections, thromboembolic events, and hospital acquired autonomy loss.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and older
* Able to provide informed consent
* ASA I and II (American Society of Anesthesiologists)
* Staying less than 50 kilometers from a hospital after surgery
* Being accompanied by an adult able to assist the patient in his recovery and to intervene in case of an emergency for the first 48 hours after surgery
* No anastomotic leak proven on preoperative water soluble enema

Exclusion Criteria:

* Language barrier or significant communication problem
* Immunosuppression
* Therapeutic anticoagulation
* Previous proctocolectomy
* Previous ileal pouch anal anastomosis
* Technical factors during surgery (conversion to midline laparotomy or other, at surgeon's discretion)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2019-06 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Total length of hospital stay | 30 days after surgery
  The number of days spent in the hospital from the time of the surgery to the time of the discharge as well as any day spent in the hospital after any readmission in the 30 days following the ileostomy closure.

SECONDARY OUTCOMES:
Readmission rate | 30 days after surgery
  Any hospitalisation after surgery
Postoperative complication rate | 30 days after surgery
  Any complication after surgery
Postoperative ileus rate | 30 days after surgery
  Ileus necessitating installation of a nasogastric tube
Postoperative surgical site infection rate | 30 days after surgery
  Infection of the surgical site
Postoperative mortality rate | 30 days after surgery
  Death after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: François Letarte, MD, MSc, Study Director — CHU de Québec-Université Laval; Xavier Paré, MD, Principal Investigator — CHU de Québec-Université Laval; Geneviève Morin, MD, Principal Investigator — CHU de Québec-Université Laval
Locations (2):
- Canada (2):
  - Hôpital Saint-François d'Assise, Québec, Quebec
  - Hôtel-Dieu de Québec, Québec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Huser N, Michalski CW, Erkan M, Schuster T, Rosenberg R, Kleeff J, Friess H. Systematic review and meta-analysis of the role of defunctioning stoma in low rectal cancer surgery. Ann Surg. 2008 Jul;248(1):52-60. doi: 10.1097/SLA.0b013e318176bf65. PMID 18580207
- [Result] Tan WS, Tang CL, Shi L, Eu KW. Meta-analysis of defunctioning stomas in low anterior resection for rectal cancer. Br J Surg. 2009 May;96(5):462-72. doi: 10.1002/bjs.6594. PMID 19358171
- [Result] Chen J, Wang DR, Yu HF, Zhao ZK, Wang LH, Li YK. Defunctioning stoma in low anterior resection for rectal cancer: a meta- analysis of five recent studies. Hepatogastroenterology. 2012 Sep;59(118):1828-31. doi: 10.5754/hge11786. PMID 22193436
- [Result] Koperna T. Cost-effectiveness of defunctioning stomas in low anterior resections for rectal cancer: a call for benchmarking. Arch Surg. 2003 Dec;138(12):1334-8; discussion 1339. doi: 10.1001/archsurg.138.12.1334. PMID 14662534
- [Result] Wong KS, Remzi FH, Gorgun E, Arrigain S, Church JM, Preen M, Fazio VW. Loop ileostomy closure after restorative proctocolectomy: outcome in 1,504 patients. Dis Colon Rectum. 2005 Feb;48(2):243-50. doi: 10.1007/s10350-004-0771-0. PMID 15714246
- [Result] D'Haeninck A, Wolthuis AM, Penninckx F, D'Hondt M, D'Hoore A. Morbidity after closure of a defunctioning loop ileostomy. Acta Chir Belg. 2011 May-Jun;111(3):136-41. doi: 10.1080/00015458.2011.11680724. PMID 21780519
- [Result] Giannakopoulos GF, Veenhof AA, van der Peet DL, Sietses C, Meijerink WJ, Cuesta MA. Morbidity and complications of protective loop ileostomy. Colorectal Dis. 2009 Jul;11(6):609-12. doi: 10.1111/j.1463-1318.2008.01690.x. Epub 2008 Oct 1. PMID 19175642
- [Result] Chow A, Tilney HS, Paraskeva P, Jeyarajah S, Zacharakis E, Purkayastha S. The morbidity surrounding reversal of defunctioning ileostomies: a systematic review of 48 studies including 6,107 cases. Int J Colorectal Dis. 2009 Jun;24(6):711-23. doi: 10.1007/s00384-009-0660-z. Epub 2009 Feb 17. PMID 19221766
- [Result] Loffler T, Rossion I, Bruckner T, Diener MK, Koch M, von Frankenberg M, Pochhammer J, Thomusch O, Kijak T, Simon T, Mihaljevic AL, Kruger M, Stein E, Prechtl G, Hodina R, Michal W, Strunk R, Henkel K, Bunse J, Jaschke G, Politt D, Heistermann HP, Fusser M, Lange C, Stamm A, Vosschulte A, Holzer R, Partecke LI, Burdzik E, Hug HM, Luntz SP, Kieser M, Buchler MW, Weitz J; HASTA Trial Group. HAnd Suture Versus STApling for Closure of Loop Ileostomy (HASTA Trial): results of a multicenter randomized trial (DRKS00000040). Ann Surg. 2012 Nov;256(5):828-35; discussion 835-6. doi: 10.1097/SLA.0b013e318272df97. PMID 23095628
- [Result] Luglio G, Pendlimari R, Holubar SD, Cima RR, Nelson H. Loop ileostomy reversal after colon and rectal surgery: a single institutional 5-year experience in 944 patients. Arch Surg. 2011 Oct;146(10):1191-6. doi: 10.1001/archsurg.2011.234. PMID 22006879
- [Result] Hiranyakas A, Rather A, da Silva G, Weiss EG, Wexner SD. Loop ileostomy closure after laparoscopic versus open surgery: is there a difference? Surg Endosc. 2013 Jan;27(1):90-4. doi: 10.1007/s00464-012-2422-1. Epub 2012 Jun 30. PMID 22752281
- [Result] Mengual-Ballester M, Garcia-Marin JA, Pellicer-Franco E, Guillen-Paredes MP, Garcia-Garcia ML, Cases-Baldo MJ, Aguayo-Albasini JL. Protective ileostomy: complications and mortality associated with its closure. Rev Esp Enferm Dig. 2012 Jul;104(7):350-4. doi: 10.4321/s1130-01082012000700003. PMID 22849495
- [Result] Gong J, Guo Z, Li Y, Gu L, Zhu W, Li J, Li N. Stapled vs hand suture closure of loop ileostomy: a meta-analysis. Colorectal Dis. 2013;15(10):e561-8. doi: 10.1111/codi.12388. PMID 24033921
- [Result] Peacock O, Bhalla A, Simpson JA, Gold S, Hurst NG, Speake WJ, Tierney GM, Lund JN. Twenty-three-hour stay loop ileostomy closures: a pilot study. Tech Coloproctol. 2013 Feb;17(1):45-9. doi: 10.1007/s10151-012-0880-z. Epub 2012 Aug 31. PMID 22936588
- [Result] Peacock O, Law CI, Collins PW, Speake WJ, Lund JN, Tierney GM. Closure of loop ileostomy: potentially a daycase procedure? Tech Coloproctol. 2011 Dec;15(4):431-7. doi: 10.1007/s10151-011-0781-6. Epub 2011 Oct 28. PMID 22033543
- [Result] Baraza W, Wild J, Barber W, Brown S. Postoperative management after loop ileostomy closure: are we keeping patients in hospital too long? Ann R Coll Surg Engl. 2010 Jan;92(1):51-5. doi: 10.1308/003588410X12518836439209. PMID 20056062
- [Result] Joh YG, Lindsetmo RO, Stulberg J, Obias V, Champagne B, Delaney CP. Standardized postoperative pathway: accelerating recovery after ileostomy closure. Dis Colon Rectum. 2008 Dec;51(12):1786-9. doi: 10.1007/s10350-008-9399-9. Epub 2008 Jun 24. PMID 18575937
- [Result] Kalady MF, Fields RC, Klein S, Nielsen KC, Mantyh CR, Ludwig KA. Loop ileostomy closure at an ambulatory surgery facility: a safe and cost-effective alternative to routine hospitalization. Dis Colon Rectum. 2003 Apr;46(4):486-90. doi: 10.1007/s10350-004-6587-0. PMID 12682542
- [Result] Gatt M, Reddy BS, Mainprize KS. Day-case stoma surgery: is it feasible? Surgeon. 2007 Jun;5(3):143-7. doi: 10.1016/s1479-666x(07)80041-2. PMID 17575667
- [Result] Bhalla A, Peacock O, Tierney GM, Tou S, Hurst NG, Speake WJ, Williams JP, Lund JN. Day-case closure of ileostomy: feasible, safe and efficient. Colorectal Dis. 2015 Sep;17(9):820-3. doi: 10.1111/codi.12961. PMID 25808587
- [Result] Sajid MS, Craciunas L, Baig MK, Sains P. Systematic review and meta-analysis of published, randomized, controlled trials comparing suture anastomosis to stapled anastomosis for ileostomy closure. Tech Coloproctol. 2013 Dec;17(6):631-9. doi: 10.1007/s10151-013-1027-6. Epub 2013 May 17. PMID 23681301
- [Result] Sajid MS, Bhatti MI, Miles WF. Systematic review and meta-analysis of published randomized controlled trials comparing purse-string vs conventional linear closure of the wound following ileostomy (stoma) closure. Gastroenterol Rep (Oxf). 2015 May;3(2):156-61. doi: 10.1093/gastro/gou038. Epub 2014 Jul 10. PMID 25011379
- [Result] Bracey E, Chave H, Agombar A, Sleight S, Dukes S, Bryan S, Branagan G. Ileostomy closure in an enhanced recovery setting. Colorectal Dis. 2015 Oct;17(10):917-21. doi: 10.1111/codi.12989. PMID 25950922
- [Result] Adamina M, Kehlet H, Tomlinson GA, Senagore AJ, Delaney CP. Enhanced recovery pathways optimize health outcomes and resource utilization: a meta-analysis of randomized controlled trials in colorectal surgery. Surgery. 2011 Jun;149(6):830-40. doi: 10.1016/j.surg.2010.11.003. Epub 2011 Jan 14. PMID 21236454
- [Result] Man VC, Choi HK, Law WL, Foo DC. Morbidities after closure of ileostomy: analysis of risk factors. Int J Colorectal Dis. 2016 Jan;31(1):51-7. doi: 10.1007/s00384-015-2327-2. Epub 2015 Aug 6. PMID 26245947
- [Result] Keller DS, Swendseid B, Khan S, Delaney CP. Readmissions after ileostomy closure: cause to revisit a standardized enhanced recovery pathway? Am J Surg. 2014 Oct;208(4):650-5. doi: 10.1016/j.amjsurg.2014.05.003. Epub 2014 Jul 5. PMID 25087854
- [Result] Abrisqueta J, Abellan I, Lujan J, Hernandez Q, Parrilla P. Stimulation of the efferent limb before ileostomy closure: a randomized clinical trial. Dis Colon Rectum. 2014 Dec;57(12):1391-6. doi: 10.1097/DCR.0000000000000237. PMID 25380005
- [Result] Kaidar-Person O, Person B, Wexner SD. Complications of construction and closure of temporary loop ileostomy. J Am Coll Surg. 2005 Nov;201(5):759-73. doi: 10.1016/j.jamcollsurg.2005.06.002. Epub 2005 Sep 6. No abstract available. PMID 16256921
- [Result] Rushworth GF, Megson IL. Existing and potential therapeutic uses for N-acetylcysteine: the need for conversion to intracellular glutathione for antioxidant benefits. Pharmacol Ther. 2014 Feb;141(2):150-9. doi: 10.1016/j.pharmthera.2013.09.006. Epub 2013 Sep 28. PMID 24080471
- [Result] Sabbagh C, Cosse C, Rebibo L, Hariz H, Dhahri A, Regimbeau JM. Identifying Patients Eligible for a Short Hospital Stay After Stoma Closure. J Invest Surg. 2018 Jun;31(3):168-172. doi: 10.1080/08941939.2017.1299818. Epub 2017 Mar 31. PMID 28362132
- [Result] Hou Y, Wang L, Yi D, Ding B, Yang Z, Li J, Chen X, Qiu Y, Wu G. N-acetylcysteine reduces inflammation in the small intestine by regulating redox, EGF and TLR4 signaling. Amino Acids. 2013 Sep;45(3):513-22. doi: 10.1007/s00726-012-1295-x. Epub 2012 Apr 25. PMID 22532030
- [Result] Wang Q, Hou Y, Yi D, Wang L, Ding B, Chen X, Long M, Liu Y, Wu G. Protective effects of N-acetylcysteine on acetic acid-induced colitis in a porcine model. BMC Gastroenterol. 2013 Aug 30;13:133. doi: 10.1186/1471-230X-13-133. PMID 24001404
- [Result] Fohl AL, Johnson CE, Cober MP. Stability of extemporaneously prepared acetylcysteine 1% and 10% solutions for treatment of meconium ileus. Am J Health Syst Pharm. 2011 Jan 1;68(1):69-72. doi: 10.2146/ajhp100214. PMID 21164069
- [Result] Bokey EL, Chapuis PH, Fung C, Hughes WJ, Koorey SG, Brewer D, Newland RC. Postoperative morbidity and mortality following resection of the colon and rectum for cancer. Dis Colon Rectum. 1995 May;38(5):480-6; discussion 486-7. doi: 10.1007/BF02148847. PMID 7736878

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-06): https://cdn.clinicaltrials.gov/large-docs/22/NCT03941522/Prot_SAP_000.pdf